CLINICAL TRIAL: NCT01965704
Title: AIM 2- Prevention of Neonatal Abstinence Syndrome
Brief Title: Can Ondansetron Prevent Neonatal Abstinence Syndrome (NAS) in Babies Born to Narcotic-dependent Women
Acronym: AIM2NAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Medical Center (Other); Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, David R. Drover, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Aim 2_RO1-HD-070795-01A1; NAS2 (Other: Stanford)
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Results first posted 2022-05-10 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Narcotic Addiction; Neonatal Abstinence Syndrome
Keywords: Narcotic addiction during pregnancy; Neonatal abstinence syndrome; NAS
MeSH Terms: conditions — Narcotic-Related Disorders; Neonatal Abstinence Syndrome | interventions — Ondansetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Ondansetron (Experimental): Pregnant Women: ondansetron 8mg intravenously (IV) within 4 hours of delivery. Neonates: ondansetron 0.07 mg/kg given orally every 24 hours starting 4-8 hours after delivery, for up to 5 days (if IV line available in neonate, ondansetron 0.04 mg/kg IV every 24 hours for up to 5 days).
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): Pregnant Women: placebo given intravenously prior to delivery (volume to mimic the IV volume of the ondansetron group).
  Neonates: placebo given orally every 24 hours, starting 4-8 hours after delivery, for up to 5 days with volume to mimic the oral volume of the ondansetron group (if IV line available, placebo may be given IV).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — Pregnant women may receive a second dose of IV ondansetron if they have not delivered within 4 hours of receiving the IV study medication. 50% of the 90 mother/baby pairs will receive ondansetron; the baby will always get the same study medication as the mother.
  Other Names: Zofran
  Arms: Ondansetron
Drug: Placebo — All doses of placebo, whether IV or oral, will mimic the same volume as the ondansetron group to maintain the blind. Pregnant women may receive a second dose of IV placebo if they have not delivered within 4 hours of being given the IV study medication. 50% of the 90 mother/baby pairs will receive placebo; the baby will always receive the same study medication as the mother.
  Other Names: IV Normal saline; oral simple syrup
  Arms: Placebo

SUMMARY:
The Investigators hope to learn if they can prevent or lessen the symptoms of neonatal abstinence syndrome (NAS) in babies born to narcotic-dependent mothers by using the drug ondansetron in the mothers prior to delivery and their babies after delivery.

The study is a randomized, double-blind, placebo-controlled study with one half the mother-baby pairs to receive ondansetron and the other half of the mother-baby pairs to receive placebo. The pregnant narcotic-dependent mothers will receive an intravenous dose of study medication prior to delivery; the neonates, after their birth, will receive the same study medication the mother received every 24 hours for up to 5 days.

The Investigators will follow up with the mother-baby pairs for 10 days after study drug has stopped and one last follow up, about 30 days after stopping study drug, to learn if the baby had any symptoms of NAS in that time period.

DETAILED DESCRIPTION:
All neonates will have a screening 12-lead EKG prior to their first dose of study medication to determine if QTc prolongation is present. A repeat 12-lead EKG will be done after each dose of study medication, approximately 2-5 hours post dose; if a neonate has prolonged QTc the study drug will be stopped.

Investigators may obtain up to 9 pharmacokinetic (PK) blood samples from the neonates over 5 days when standard of care blood samples are drawn. These samples will consist of 1 to 2 drops of blood collected on filter paper and sent to Stanford for PK analysis.

The modified Finnegan scoring system will be used to evaluate neonates for symptoms of NAS at each site and it is considered standard-of-care for babies at risk of NAS. Morphine will be the first treatment choice before other treatment medication choices (opioid or non-opioid) for NAS symptoms. Each site involved has established guidelines for starting, advancing and weaning treatment for NAS. Any medication used to treat NAS will be recorded.

Interim analysis: will be performed after the first 20 pregnant women and their neonates have been enrolled and dosed with study drug. (Interim Analysis was done on first 21 mother/baby pairs in May 2016).

To protect the confidentiality of the patients (study subjects), the lead site, Stanford University, received a Certificate of Confidentiality from the NIH.

ELIGIBILITY:
Inclusion Criteria:

* adult female, opioid-dependent for at least 3 weeks prior to delivery.
* adult female, otherwise healthy.
* adult female, age 18-45 years inclusive.
* adult female, signed consent to participate for self and neonate (maternal subject may decide not to receive the study drug but her neonate can still be included in the study).
* neonate, gestational age 37 weeks through 41 weeks and 6 days at birth.
* neonate, corrected QT interval (QTc) from 12-lead electrocardiogram (ECG) less than 480 milliseconds (ms).

Exclusion Criteria:

* adult female, any condition that, in the opinion of the investigator, would compromise the health of the participant (both mother and fetus) or the integrity of the data.
* adult female, known allergy to study drug (ondansetron).
* adult female, screening 12-lead ECG, if done, showing prolonged QTc will stop the mother from receiving any study drug but her neonate can still be included in the study.
* adult female, not dependent on opioids for at least 3 weeks prior to delivery.
* adult female, generally not healthy.
* adult female, age 17 years or less or 46 years of age and older.
* adult female and neonate, the maternal ingestion or administration of ondansetron within 24 hours prior to delivery, for reasons other than study purposes, will exclude the mother and the neonate.
* neonate, preterm or post-term gestational age at delivery.
* neonate, QTc showing results greater than or equal to 480ms on any 12-lead ECG post delivery will stop the dosing of the study drug, but safety follow up will be done if the mother or baby received at least one dose of study drug.

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 196 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Drover, MD, Principal Investigator — Stanford University
Locations (8):
- United States (8):
  - UCSF, San Francisco General Hospital, San Francisco, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Stanford University Medical Center, Stanford, California
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - The University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
We will not share any individual participant data with other researchers.

REFERENCES:
- [Derived] Peltz G, Jansson LM, Adeniyi-Jones S, Cohane C, Drover D, Shafer S, Wang M, Wu M, Govindaswami B, Jegatheesan P, Argani C, Khan S, Kraft WK. Ondansetron to reduce neonatal opioid withdrawal severity a randomized clinical trial. J Perinatol. 2023 Mar;43(3):271-276. doi: 10.1038/s41372-022-01487-2. Epub 2022 Aug 27. PMID 36030327

RESULTS

PARTICIPANT FLOW:
Groups:
- Ondansetron - Mothers: Pregnant Women: ondansetron 8mg intravenously (IV) within 4 hours of delivery; may receive a second dose of IV ondansetron if they have not delivered within 4 hours of receiving the IV study medication.
- Ondansetron - Neonates: Neonates: ondansetron 0.07 mg/kg given orally every 24 hours starting 4-8 hours after delivery, for up to 5 days (if IV line available in neonate, ondansetron 0.04 mg/kg IV every 24 hours for up to 5 days).
- Placebo - Mothers: Pregnant Women: placebo given intravenously prior to delivery (volume to mimic the IV volume of the ondansetron group); may receive a second dose of IV placebo if they have not delivered within 4 hours of being given the IV study medication.
- Placebo - Neonates: Neonates: placebo given orally every 24 hours, starting 4-8 hours after delivery, for up to 5 days with volume to mimic the oral volume of the ondansetron group (if IV line available, placebo may be given IV).
Period: Overall Study
Arm/Group | Ondansetron - Mothers | Ondansetron - Neonates | Placebo - Mothers | Placebo - Neonates
Started | 48 | 48 | 50 | 50
Received Intervention | 45 | 45 | 47 | 47
Analyzable Population (Received treatment and met all eligibility criteria) | 45 | 45 | 41 | 41
Completed | 45 | 45 | 45 | 45
Not Completed | 3 | 3 | 5 | 5
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 1
Not completed — Delivered at home | 1 | 1 | 0 | 0
Not completed — Experienced complications | 0 | 0 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Did not meet inclusion criteria | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol and met all inclusion criteria are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ondansetron - Mothers | Ondansetron - Neonates | Placebo - Mothers | Placebo - Neonates | Total
Number analyzed (Participants) | 45 | 45 | 41 | 41 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 45 | 0 | 41 | 86
  Between 18 and 65 years | 45 | 0 | 41 | 0 | 86
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 22 | 41 | 19 | 127
  Male | 0 | 23 | 0 | 22 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 4 | 4 | 20
  White | 35 | 35 | 34 | 34 | 138
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 3 | 3 | 3 | 3 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 45 | 41 | 41 | 172
Gestational age at birth [Median (Full Range); unit: weeks] — Population: Gestational age at birth was assessed in the neonates only.
  weeks
    number analyzed (Participants) | 0 | 45 | 0 | 41 | 86
    (all) |  | 39 [36 to 41] |  | 39 [37 to 40] | 39 [36 to 41]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Neonatal Abstinence Syndrome
Description: The incidence of neonatal abstinence syndrome (NAS) measured as the number of neonates who need for morphine treatment for the symptoms of neonatal opioid withdrawal syndrome (NOWS) while the neonates received study medication and for the 30 days after stopping the study medication.
Time Frame: 35 days
Population: Neonates who completed the protocol and met all inclusion criteria are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ondansetron - Neonates | Placebo - Neonates
Number analyzed (Participants) | 45 | 41
Participants | 22 | 26
Statistical Analysis 1: Comparison: Ondansetron - Neonates vs Placebo - Neonates; Test type: Other; p = 0.2, Fisher Exact

2. Secondary Outcome: Length of Hospital Stay
Description: Severity of NAS will be measured by neonates' length of hospital stay (birth to discharge). Length of stay was calculated with 1) no maximum length, and 2) maximum length of stay capped at 15 days. All participants were included in both analyses.
Time Frame: At Day 15 and up to 64 days
Population: Neonates who completed the protocol and met all inclusion criteria are included in the analysis.
Measure: Mean (Full Range); unit: days
Arm/Group | Ondansetron - Neonates | Placebo - Neonates
Number analyzed (Participants) | 45 | 41
days
  Mean hospital stay | 15.5 [2 to 64] | 17.4 [3 to 63]
  Mean hospital stay with a 15-day maximum | 9.3 [2 to 15] | 11.2 [3 to 15]
Statistical Analysis 1: Comparison: Ondansetron - Neonates vs Placebo - Neonates; Difference in overall length of stay; Test type: Other; p = 0.56, Wilcoxon Rank-Sum test; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-8.0 to 4.3] — The 95% confidence interval between the ondansetron group and the placebo group was calculated with the use of Hodges-Lehmann estimator
Statistical Analysis 2: Comparison: Ondansetron - Neonates vs Placebo - Neonates; Difference in length of stay as calculated with maximum length capped at 15 days; Test type: Other; p = 0.07, Wilcoxon Rank-Sum test; Median Difference (Final Values) = -1.9, 95% CI 2-sided [-4.0 to 0.2] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Total Dose of Narcotic Required to Treat the Symptoms of NAS
Description: Median dose of morphine required by neonates within 15 days of delivery.
Time Frame: 15 days
Population: Neonates who completed the protocol and met all inclusion criteria are included in the analysis.
Measure: Median (Full Range); unit: mg
Arm/Group | Ondansetron - Neonates | Placebo - Neonates
Number analyzed (Participants) | 45 | 41
mg | 9.3 [0.8 to 37.4] | 11.1 [0.8 to 31.1]
Statistical Analysis 1: Comparison: Ondansetron - Neonates vs Placebo - Neonates; Test type: Other; p = 0.31, Wilcoxon Rank-Sum test; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-8.8 to 2.7] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Participants Requiring Adjunctive Medication to Treat NOWS
Description: Number of neonates requiring treatment with phenobarbital or clonidine.
Time Frame: 15 days
Population: Neonates who completed the protocol and met all inclusion criteria are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ondansetron - Neonates | Placebo - Neonates
Number analyzed (Participants) | 45 | 41
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | Ondansetron - Mothers | Ondansetron - Neonates | Placebo - Mothers | Placebo - Neonates
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/48 | 2/48 | 1/50 | 4/50
Other Adverse Events (participants affected / at risk) | 1/48 | 18/48 | 1/50 | 15/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ondansetron - Mothers (N=48) | Ondansetron - Neonates (N=48) | Placebo - Mothers (N=50) | Placebo - Neonates (N=50)
Hypoxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 — Brain injury related to low oxygen at birth
Readmission for NOWS observation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
C-section superficial wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Late onset NOWS (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intermittent seizures (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ondansetron - Mothers (N=48) | Ondansetron - Neonates (N=48) | Placebo - Mothers (N=50) | Placebo - Neonates (N=50)
Subcutaneous hematoma drainage from C-section incision (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Vaginal bleeding (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Prolonged QTc interval (Cardiac disorders) | 0 | 14 | 0 | 12
Short QTc interval (Cardiac disorders) | 0 | 3 | 0 | 2
Cyanotic episode (Cardiac disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Laryngomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Left brachial plexus injury (Nervous system disorders) | 0 | 0 | 0 | 1
Secundum atrial septal defect (Cardiac disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2019-03-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT01965704/Prot_002.pdf
  • Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT01965704/SAP_003.pdf
  • Informed Consent Form: Parental Permission (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT01965704/ICF_000.pdf
  • Informed Consent Form: Maternal ICF (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT01965704/ICF_001.pdf